CLINICAL TRIAL: NCT00457782
Title: A Phase I, Open-Label, Dose-escalation, Multicentre Study of KW-2478 Administered as a Single Agent Intravenously in a Consecutive Dosing Schedule in Patients With Relapsed/Refractory Multiple Myeloma, Chronic Lymphocytic Leukaemia or B-cell Non-Hodgkin's Lymphoma
Brief Title: A Phase I Safety, PK and PD Study of KW-2478 in Patients With Multiple Myeloma, Chronic Lymphocytic Leukaemia or B-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin UK, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2478-EU-001
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Multiple Myeloma; Chronic Lymphocytic Leukaemia; B-cell Non-Hodgkin's Lymphoma
Keywords: Cancer; Blood disorders; Leukaemia, Adult Chronic; Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Leukemia, B-Cell; Lymphoma, B-Cell; Neoplasms; Hematologic Diseases; Leukemia; Bronchiolitis Obliterans Syndrome; Lymphoma | interventions — KW-2478

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): Intravenous KW-2478 (ascending dose cohorts)
  Interventions: Drug: KW-2478

INTERVENTIONS:
Drug: KW-2478 — Daily intravenous KW-2478 for 5 days in 14-day cycles, ascending dose cohorts

SUMMARY:
The aim of this study is to determine the safety, tolerability and dose-limiting toxicities of KW-2478 and to determine the Maximum Tolerated Dose and recommended Phase II dose for patients with relapsed/refractory MM, CLL or B-cell NHL.

DETAILED DESCRIPTION:
This is a Phase I, open-label, dose-escalation study of KW-2478 in patients with relapsed/refractory multiple myeloma, chronic lymphocytic leukaemia or B-cell Non-Hodgkin's lymphoma who have no established therapeutic alternatives. Up to 42 patients will be enrolled at up to six investigational sites over a period of approximately 12 months until an MTD is reached. An additional 12 patients may be enrolled at the MTD in an expanded cohort of one or more of the eligible conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of Multiple Myeloma, Chronic Lymphocytic Leukaemia, or B-cell Non-Hodgkin's Lymphoma, who have had at least two prior standard treatment regimens and are without established therapeutic alternatives.
2. Signed IEC-approved informed consent
3. ECOG performance status of 0, 1 or 2;
4. Life expectancy of at least 3 months;
5. Adequate haematologic status, liver function and renal function
6. Patients of reproductive potential must agree to follow accepted birth control methods during the study

Exclusion Criteria:

1. No anti-cancer treatment for ≥ 3 weeks prior to receiving study drug
2. Any other severe, acute or chronic illness
3. No other prior or concurrent malignancy
4. Immunosuppressant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-04; Primary Completion 2010-08 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To determine Safety & Tolerability by adverse event rates in order to determine recommended Phase II dose | At every visit and at the end of each 14-day treatment cycle

SECONDARY OUTCOMES:
Pharmacokinetics and Pharmacodynamics | At baseline and steady state during cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Responsible Medical Officer KHKUK, Study Director — Kyowa Hakko Kirin UK; J D Cavenagh, MD. MRCP, MRCPath, Principal Investigator — St Bartholomew's Hospital, London, UK
Locations (6):
- United Kingdom (6):
  - St Bartholomew's Hospital, London
  - UCLH, London
  - Christie Hospital, Manchester
  - Nottingham University NHS Trust, Nottingham
  - Cancer Research UK Clinical Centre, Southampton
  - Royal Marsden Hospital, Sutton